CLINICAL TRIAL: NCT04521868
Title: A 6-month Study to Evaluate Sulforaphane add-on Effects in Treatment of Negative Symptoms and Cognition Impairment of Schizophrenia Patients
Brief Title: A 6-month Study to Evaluate Sulforaphane Effects in Schizophrenia Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Renrong Wu, Professor, Central South University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Jiangyin-Sulforaphane
Record Dates: First submitted 2020-08-18; First posted 2020-08-21 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Schizophrenia
Keywords: schizophrenia; sulforaphane
MeSH Terms: conditions — Schizophrenia | interventions — sulforaphane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants and researchers are blind to treatment allocation (double-blind). An independent researcher developed the computer-generated randomization plan.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- sulforaphane (Experimental): The goal of the study is to investigate whether adding sulforaphane will benefit the negative symptoms and cognitive function in individuals who have schizophrenia.
  Interventions: Drug: Sulforaphane
- placebo (Placebo Comparator): The purpose of including placebo is to judge if the outcome is related to the study medication rather than other reasons.
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Drug: Sulforaphane — Sulforaphane is a compound that can be extracted from broccoli, Brussel sprouts, cabbage, and other cruciferous plants.
  Other Names: Nutramax
  Arms: sulforaphane
Dietary Supplement: placebo — Placebo is made of starch
  Arms: placebo

SUMMARY:
The goal of the study is to investigate whether adding sulforaphane will benefit the negative symptoms and cognitive function in individuals who have schizophrenia.

This study will compare the sulforaphane with placebo. There is a thirty percent change (less than half) of receiving the placebo. The purpose of including placebo is to judge if the outcome is related to the study medication rather than other reasons.

DETAILED DESCRIPTION:
This study will be carried out in The Third Jiangyin Hospital in China and total of 120 schizophrenia patients with one negative symptom item score of PANSS≥3 will be enrolled into the study. Individuals who participate in the study will be followed for 24 weeks. The changes in clinical symptoms and neurocognitive function will be assessed from baseline (week-0) to week-12, and week-24.

ELIGIBILITY:
Inclusion Criteria:

1. Meet The Diagnostic and Statistical Manual (DSM-5) diagnostic criteria for schizophrenia;
2. First onset or duration of illness less than 30 years with current symptoms in a stable condition;
3. Male and female aged 18 to 50 years;
4. Total score greater than or equal to 20 on the sum of the seven items constituting the Positive and Negative Syndrome Scale (PANSS) negative symptoms; an item of PANSS negative symptoms >3 scores;
5. Signed the study consent for participation.

Exclusion Criteria:

1. has a history of substance dependence or abuse or whose symptoms are caused by other diagnosable mental disorders;
2. has a history of traumatic brain injury, seizures, or other known neurological diseases of the central nervous system;
3. taking antidepressants, stimulants, mood stabilizers, or received modified electroconvulsive therapy (MECT) or rTMS during the past three months;
4. having current suicidal or homicidal thoughts or any safety concern by research staff that cannot be managed during the trial;
5. taking dementia-related drugs, minocycline, and other drugs that may affect cognitive function;
6. Laboratory tests indicated significant abnormalities in blood routine, liver and kidney function, or other metabolic results;
7. pregnant or lactating women.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 125 (Actual)
Dates: Start 2020-08-31 (Actual); Primary Completion 2022-08-12 (Actual); Study Completion 2022-08-12 (Actual)

PRIMARY OUTCOMES:
Change of clinical symptoms by PANSS | 24 weeks
  The change of Positive And Negative Syndrome Scale (PANSS) total, positive and negative symptoms before and after treatment at different follow up point. The PANSS total score ranges from 30-210 points,the higher the score, the worse the symptoms.
Cognitive improvement assessed using the MATRICS Consensus Cognitive Battery (MCCB) composite score | 24 weeks
  The investigators will use the MATRICS Consensus Cognitive Battery (MCCB) Composite score as primary cognitive outcome measure.The MCCB total score is about 50 in healthy participants, patients with schizophrenia are reported to have scores as low as two standard deviations below the mean points; the higher the score, the better the cognition performance.

SECONDARY OUTCOMES:
side effects by TESS | 24 weeks
  The investigators will evaluate side effect by Treatment Emergent Symptom Scale. It is consisted of behavioural toxicity, laboratory abnormalities, nervous system, automatic nervous system, cardiovascular system and six other aspects, was used to evaluate adverse drug reactions based on the scores, ranging from 0 to 4 (the higher the score, the more serious the adverse reactions).
Change of clinical symptoms by SANS | 24 weeks
  The change of Scale for Assessment of Negative Symptoms (SANS) to evaluate negative symptoms before and after treatment at different time point. It measures 25 items of negative symptoms across 5 categories: affective blunting, alogia, avolition-apathy, anhedonia-asociality, and inattention, ranging from 0-120.
Change of clinical symptoms of CGI | 24 weeks
  The change of Clinical Global Impression (CGI) before and after treatment at different follow up point. Its assess Severity of Illness (CGI-S), Global Improvement (CGI-I), and Efficacy Index (CGI-E). CGI-S is a 7-point scale, the higher score means the more severe the illness; CGI-I is a 7 point scale, the higher score means the less improved symptoms after treatment; CGI-E is is a 4×4 rating scale that assesses the therapeutic effect of treatment with psychiatric medication and associated side effects.
Change of psychological, social, and occupational functioning by GAF | 24 weeks
  The change of Global Assessment of Functioning (GAF) Scale before and after treatment at different follow up point.ranging from 0 to 100.The higher scores means the better functioning performance.

CONTACTS AND LOCATIONS:
Overall Officials: Renrong Wu, M.D Ph.D, Principal Investigator — Central South University
Locations (1):
- Second Xiangya Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Huang J, Chen A, Jin H, Liu F, Hei G, Teng Z, Xiao J, Wu R, Zhao J, Davis JM, Shao P, Smith RC. Efficacy and Safety of Sulforaphane Added to Antipsychotics for the Treatment of Negative Symptoms of Schizophrenia: A Randomized Controlled Trial. J Clin Psychiatry. 2025 Jan 20;86(1):24m15272. doi: 10.4088/JCP.24m15272. PMID 39832347